CLINICAL TRIAL: NCT06369493
Title: The Interaction of The Gingival And Tooth Morphometric Parameters On The Gingival Phenotype
Brief Title: Examining The Relationship Between Gingival Thickness and Tooth and Gingival Parameters
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sude Yildirim, Research Assistant, Ondokuz Mayıs University
Other Study IDs: OMUKAEK: 2022/210
Record Dates: First submitted 2024-04-01; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Gingival Thickness
Keywords: Gingival Phenotype; gingival thickness; periodontium; crown morphology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thin Gingival Phenotype: Thin phenotype group: Gingival thickness ≤1 mm
- Thick Phenotype: Thick phenotype group: Gingival thickness > 1 mm

SUMMARY:
This study aims to assess whether there is a valid correlation between the identified multiple clinical and morphometric parameters and the gingival thickness.

DETAILED DESCRIPTION:
This study focused on the relationship between the clinical parameters of crown and gingival morphology and gingival phenotypes. This study investigated the relationship between clinical and morphological parameters and gingival phenotype and included all teeth up to the first molar. It also compares gingival phenotypes across arch locations and tooth groups.

Study Design and Participants:

This was a cross-sectional, controlled, randomized, and analytical data study.

This cross-sectional study was conducted with 50 participants (21 females, 29 males) aged 18-31 (mean age 22.42 ± 2.87 years) who applied to the Ondokuz Mayis University Faculty of Dentistry's Periodontology Department for periodontal treatment between September 2022 and May 2023. The statistical power of the study based on crown morphology was determined to be 80%, with a type 1 error rate of 0.05, and a sample size of at least 42 people was determined. The study was conducted in accordance with the principles of the Helsinki Declaration and with the approval of the Ondokuz Mayis University Clinical Research Ethics Committee (OMUKAEK-Protocol No:2022/210. All participants provided written informed consent prior to enrollment.

Fifty participants were divided into two groups based on the GT measurement taken from the point corresponding to the base of the gingival sulcus and categorized as thin (GT:≤ 1 mm) and thick (GT: &amp;amp;gt; 1 mm).

Clinic Measurements

Clinical periodontal parameters, including Plaque Index (PI), Gingival Index (GI), Bleeding on Probing Index (BPI), and probing pocket depth in six regions (mesial labial, midfacial, distal labial, mesial palatal, midpalatal and distal palatal) of each tooth with University of North Carolina (UNC) probe.

To reduce pain before the direct measurement, xylocaine spray (10% lidocaine) was applied. GT was measured by with a 20-gauge endodontic file in the buccal region of the incisors, canines, premolars, and first molars in both the upper and lower jaws, corresponding to the base of the gingival sulcus. After fixing the plastic stopper, the distance between the stopper and the tip of the endodontic file was measured using a modified digital caliper with 0.01 mm precision.

Papilla Length (PL) was determined by measuring the distance between the zenith points of adjacent teeth and the perpendicular line connecting to the apex of the papilla with a periodontal probe. Each tooth position had its mesial PL recorded.

The functional method proposed by Olssoni et al. was used to measure the keratinized gingival width (KGW). KGW was measured to the nearest 0.5 mm from the marginal gingiva&amp;amp;#39;s mid-buccal position to the mucogingival junction.

Measurements of Dental Stone Models

An alginate impression of the upper and lower jaw was taken in a stock tray and poured in Type 3 hard plaster according to the manufacturer's specifications to obtain the study model. The following assessments were made on the casts using a digital caliper according to the recommendations of Olssoni et al.

Crown length (CL) was determined by measuring the distance between the gingival margin or, if discernible, the cemento-enamel junction and the incisal edge of the crown. the crown.

Crown width (CW) was determined by dividing the length of the crown into three portions of equal-height; cervical (C), middle (M), and incisal (I). The distance between the approximal tooth surfaces was measured at the border between portions C and M.

Following these measurements, the ratio of crown width (CW)/ crown length (CL) was calculated for each tooth.

Using a digital angle gauge with a measurement range of 0-999.9º and a precision of 0.3º, the gingival angle (GA) was calculated by connecting the angle between two lines at the most apical part of the gingival margin of each measured tooth and the most coronal parts of the two adjacent papillae.

Intra-Examiner Repeatability:

All measurements were performed by a single examiner (SY), and intra-examiner reliability was assessed by repeating the GT measurements on 10 randomly selected participants 2 weeks later.

Statistical Analysis

Statistical analyses were performed using a statistical software package. Spearman's Correlation analysis was used to examine the relationship between parameters that did not follow a normal distribution. Binary Logistic Regression Analysis was used to examine the parameters related to gingival thickness. receiver operating characteristic (ROC) analysis was used to determine the cut-off values for parameters in predicting gingival thickness. To assess the consistency of repeated measurements by the researcher, the intraclass correlation coefficient (ICC) was used. Statistical significance level was considered p&amp;amp;lt; 0.05 Data are expressed as means ± standard deviations and median (minimum-maximum).

The relationship and interaction of clinical and morphometric parameters were recorded on the basis of individuals, tooth groups, and dental arch location.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers ≥18 years old
* Periodontal health with ≤10% bleeding on full mouth probing.
* Participants with no history of systemic diseases or consistent medication use.
* Participants with teeth present in the maxillary and mandibular anterior and posterior regions, with a measured clinical attachment level (CAL) ≤ 3 mm; without buccal attachment loss or gingival inflammation
* Participants with no evidence of dental caries, crown shape alterations, or restorations affecting the occlusal edge in the maxillary and mandibular teeth, and no radiographic evidence of bone loss
* At least one tooth in maxillary and mandibular segments, representing molar and premolar regions
* No tooth loss due to periodontal reasons

Exclusion Criteria:

* Pregnant or lactating women
* Participants who have received or are receiving orthodontic treatment and using removable dentures or orthodontic devices
* Participants with a history of periodontitis or periodontal surgery involving teeth
* Presence of abrasion or erosion in teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants applying to Ondokuz Mayis University Department of Periodontology
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Evaluation of the correlation between KGW, CW, CL PH parameters of GT measured in "mm" with a digital caliper with 0.001 mm precision in 1200 teeth in 50 participants using Spearman correlation analysis. | 1 month
  Spearman Correlation Analysis is a statistical technique in evaluating the correlation between clinical and morphometric parameters and is used to evaluate the relationship between variables. Variables GT, KGW, PH, CW, CL in 1200 teeth of 50 participants were measured in "mm" with a digital caliper with a precision of 0.001 mm. Spearman correlation coefficient takes a value between -1 and +1. +1 indicates a perfect positive monotonic relationship, -1 indicates a perfect negative monotonic relationship, and 0 indicates no relationship.
Evaluation of the effect of GT on keratinized gingival width, measured in "mm" by digital caliper with a precision of 0.001 mm, both by binary logistic regression analysis of 50 participants. | From September 2022 to May 2023
  In this study, GT, KGW are parametric variables and were measured in mm with a digital caliper with a precision of 0.001 mm. Binary logistic regression analysis is a statistical technique used to model the relationship of a dependent variable between two categorical classes. A significant p-value (<0.05) indicates that the independent variable (GT for this study) has a significant effect in the model. Binary logistic regression analysis expresses the effect of independent variables on the dependent variable in terms of log-odds. The coefficients of the model determine the magnitude and direction of the effect of the independent variables.
Examining the effect of age and gender of 50 participants on the gingival thickness measured in mm using binary logistic regression analysis. | 1 month
  In this study, GT is a parametric variable and is measured in mm. The effect of age and gender on GT of 50 participants over the age of 18 was examined with binary logistic regression analysis. Binary logistic regression analysis is a statistical technique used to model the relationship of a dependent variable between two categorical classes. A significant p value (<0.05) indicates that the independent variable (GT for this study) has a significant effect in the model. Binary logistic regression analysis expresses the effect of independent variables on the dependent variable in log-odds terms. The coefficients of the model determine the magnitude and direction of the effect of the independent variables.

OTHER OUTCOMES:
Evaluation of researcher reliability by ICC (Intra-Class Correlation Coefficient) in 10 participants in 2 weeks | Baseline to 2 weeks
  ICC (Intraclass Correlation Coefficient) is a statistical measure used to evaluate the reliability of repeated measurements or observations. The ICC value varies between 0 and 1. An ICC value approaching 1 indicates perfect agreement between measurements, while an ICC value approaching 0 indicates discordance or inconsistency between measurements. In this study, gingival thickness measurements in 10 participants were measured again by the same researcher at 2-week intervals to investigate their reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University Faculty of Dentistry Department of Periodonthology, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolte R, Kolte A, Mahajan A. Assessment of gingival thickness with regards to age, gender and arch location. J Indian Soc Periodontol. 2014 Jul;18(4):478-81. doi: 10.4103/0972-124X.138699. PMID 25210263
- [Background] Yin XJ, Wei BY, Ke XP, Zhang T, Jiang MY, Luo XY, Sun HQ. Correlation between clinical parameters of crown and gingival morphology of anterior teeth and periodontal biotypes. BMC Oral Health. 2020 Feb 19;20(1):59. doi: 10.1186/s12903-020-1040-x. PMID 32075626
- [Background] Chou YH, Tsai CC, Wang JC, Ho YP, Ho KY, Tseng CC. New classification of crown forms and gingival characteristics in taiwanese. Open Dent J. 2008 Nov 28;2:114-9. doi: 10.2174/1874210600802010114. PMID 19444325
- [Background] Vlachodimou E, Fragkioudakis I, Vouros I. Is There an Association between the Gingival Phenotype and the Width of Keratinized Gingiva? A Systematic Review. Dent J (Basel). 2021 Mar 23;9(3):34. doi: 10.3390/dj9030034. PMID 33806934
- [Background] Chow YC, Eber RM, Tsao YP, Shotwell JL, Wang HL. Factors associated with the appearance of gingival papillae. J Clin Periodontol. 2010 Aug 1;37(8):719-27. doi: 10.1111/j.1600-051X.2010.01594.x. Epub 2010 Jul 1. PMID 20618545
- [Background] AlQahtani NA, Haralur SB, AlMaqbol M, AlMufarrij AJ, Al Dera AA, Al-Qarni M. Distribution of smile line, gingival angle and tooth shape among the Saudi Arabian subpopulation and their association with gingival biotype. J Int Soc Prev Community Dent. 2016 Apr;6(Suppl 1):S53-8. doi: 10.4103/2231-0762.181168. PMID 27195228
- [Background] Fischer KR, Richter T, Kebschull M, Petersen N, Fickl S. On the relationship between gingival biotypes and gingival thickness in young Caucasians. Clin Oral Implants Res. 2015 Aug;26(8):865-869. doi: 10.1111/clr.12356. Epub 2014 Mar 1. PMID 24580810
- [Background] Collins JR, Pannuti CM, Veras K, Ogando G, Brache M. Gingival phenotype and its relationship with different clinical parameters: a study in a Dominican adult sample. Clin Oral Investig. 2021 Aug;25(8):4967-4973. doi: 10.1007/s00784-021-03806-x. Epub 2021 Jan 29. PMID 33515119
- [Background] Olsson M, Lindhe J, Marinello CP. On the relationship between crown form and clinical features of the gingiva in adolescents. J Clin Periodontol. 1993 Sep;20(8):570-7. doi: 10.1111/j.1600-051x.1993.tb00773.x. PMID 7691897
- [Background] Muller HP, Kononen E. Variance components of gingival thickness. J Periodontal Res. 2005 Jun;40(3):239-44. doi: 10.1111/j.1600-0765.2005.00798.x. PMID 15853970
- [Background] Vandana KL, Savitha B. Thickness of gingiva in association with age, gender and dental arch location. J Clin Periodontol. 2005 Jul;32(7):828-30. doi: 10.1111/j.1600-051X.2005.00757.x. PMID 15966893
- [Background] Fischer KR, Buchel J, Kauffmann F, Heumann C, Friedmann A, Schmidlin PR. Gingival phenotype distribution in young Caucasian women and men - An investigative study. Clin Exp Dent Res. 2022 Feb;8(1):374-379. doi: 10.1002/cre2.482. Epub 2021 Nov 11. PMID 34766469
- [Background] Kim DM, Bassir SH, Nguyen TT. Effect of gingival phenotype on the maintenance of periodontal health: An American Academy of Periodontology best evidence review. J Periodontol. 2020 Mar;91(3):311-338. doi: 10.1002/JPER.19-0337. Epub 2020 Jan 16. PMID 31691970
- [Background] Shao Y, Yin L, Gu J, Wang D, Lu W, Sun Y. Assessment of Periodontal Biotype in a Young Chinese Population using Different Measurement Methods. Sci Rep. 2018 Jul 25;8(1):11212. doi: 10.1038/s41598-018-29542-z. PMID 30046153
- [Background] La Rocca AP, Alemany AS, Levi P Jr, Juan MV, Molina JN, Weisgold AS. Anterior maxillary and mandibular biotype: relationship between gingival thickness and width with respect to underlying bone thickness. Implant Dent. 2012 Dec;21(6):507-15. doi: 10.1097/ID.0b013e318271d487. PMID 23147165
- [Background] undefined
- [Background] Fischer KR, Kunzlberger A, Donos N, Fickl S, Friedmann A. Gingival biotype revisited-novel classification and assessment tool. Clin Oral Investig. 2018 Jan;22(1):443-448. doi: 10.1007/s00784-017-2131-1. Epub 2017 May 27. PMID 28551728
- [Background] Shah R, Sowmya NK, Mehta DS. Prevalence of gingival biotype and its relationship to clinical parameters. Contemp Clin Dent. 2015 Sep;6(Suppl 1):S167-71. doi: 10.4103/0976-237X.166824. PMID 26604569
- [Background] Olsson M, Lindhe J. Periodontal characteristics in individuals with varying form of the upper central incisors. J Clin Periodontol. 1991 Jan;18(1):78-82. doi: 10.1111/j.1600-051x.1991.tb01124.x. PMID 2045523
- [Background] Fischer KR, Grill E, Jockel-Schneider Y, Bechtold M, Schlagenhauf U, Fickl S. On the relationship between gingival biotypes and supracrestal gingival height, crown form and papilla height. Clin Oral Implants Res. 2014 Aug;25(8):894-8. doi: 10.1111/clr.12196. Epub 2013 May 30. PMID 23718206
- [Background] Stellini E, Comuzzi L, Mazzocco F, Parente N, Gobbato L. Relationships between different tooth shapes and patient's periodontal phenotype. J Periodontal Res. 2013 Oct;48(5):657-62. doi: 10.1111/jre.12057. Epub 2013 Feb 27. PMID 23441885
- [Background] Joshi A, Suragimath G, Zope SA, Ashwinirani SR, Varma SA. Comparison of Gingival Biotype between different Genders based on Measurement of Dentopapillary Complex. J Clin Diagn Res. 2017 Sep;11(9):ZC40-ZC45. doi: 10.7860/JCDR/2017/30144.10575. Epub 2017 Sep 1. PMID 29207831
- [Background] Stein JM, Lintel-Hoping N, Hammacher C, Kasaj A, Tamm M, Hanisch O. The gingival biotype: measurement of soft and hard tissue dimensions - a radiographic morphometric study. J Clin Periodontol. 2013 Dec;40(12):1132-9. doi: 10.1111/jcpe.12169. Epub 2013 Oct 16. PMID 24102580
- [Background] De Rouck T, Eghbali R, Collys K, De Bruyn H, Cosyn J. The gingival biotype revisited: transparency of the periodontal probe through the gingival margin as a method to discriminate thin from thick gingiva. J Clin Periodontol. 2009 May;36(5):428-33. doi: 10.1111/j.1600-051X.2009.01398.x. PMID 19419444
- [Background] Belak S, Zizka R, Starosta M, Zapletalova J, Sedy J, Stefanatny M. The influence of gingival phenotype on the morphology of the maxillary central papilla. BMC Oral Health. 2021 Jan 23;21(1):43. doi: 10.1186/s12903-021-01400-x. PMID 33485351
- [Derived] Bolat SY, Guliyev R, Lutfioglu M. A comprehensive analysis of gingival phenotype: interaction and relationship between gingival and tooth morphometric parameters. BMC Oral Health. 2025 Sep 26;25(1):1450. doi: 10.1186/s12903-025-06821-6. PMID 41013551